CLINICAL TRIAL: NCT02924688
Title: A Phase III, Randomized, Double-blind, Active Controlled, Parallel Group Study, Comparing the Efficacy, Safety and Tolerability of the Fixed Dose Combination FF/UMEC/VI With the Fixed Dose Dual Combination of FF/VI, Administered Once-daily Via a Dry Powder Inhaler in Subjects With Inadequately Controlled Asthma
Brief Title: A Phase III Parallel Group Study, Comparing the Efficacy, Safety and Tolerability of the Fixed Dose Combination (FDC) of Fluticasone Furoate+Umeclidinium Bromide+Vilanterol (FF/UMEC/VI) With the FDC of FF/VI in Subjects With Inadequately Controlled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205715; 2016-001304-37 (EudraCT Number)
Record Dates: First submitted 2016-09-12; First posted 2016-10-05 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: umeclidinium bromide; fluticasone furoate; vilanterol; fixed dose combination; lung function; albuterol/salbutamol; asthma; closed triple therapy
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Albuterol; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- FF/UMEC/VI (100/31.25/25) mcg closed triple therapy (Experimental): Subjects will receive FF/UMEC/VI (100/31.25/25) mcg inhalation powder via DPI, once daily in the morning. Subjects may receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/UMEC/VI (100/31.25/25) mcg; Drug: FF/VI (100/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)
- FF/UMEC/VI (100/62.5/25) mcg closed triple therapy (Experimental): Subjects will receive FF/UMEC/VI (100/62.5/25) mcg inhalation powder via DPI, once daily in the morning. Subjects will also receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/UMEC/VI (100/62.5/25) mcg; Drug: FF/VI (100/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)
- FF/UMEC/VI (200/31.25/25) mcg closed triple therapy (Experimental): Subjects will receive FF/UMEC/VI (200/31.25/25) mcg inhalation powder via DPI, once daily in the morning. Subjects may receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/UMEC/VI (200/31.25/25) mcg; Drug: FF/VI (100/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)
- FF/UMEC/VI (200/62.5/25) mcg closed triple therapy (Experimental): Subjects may receive FF/UMEC/VI (200/62.5/25) mcg inhalation powder via DPI, once daily in the morning. Subjects may receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/UMEC/VI (200/62.5/25) mcg; Drug: FF/VI (100/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)
- FF/VI (100/25) mcg dual combination therapy (Active Comparator): Subjects will receive FF/VI (100/25) mcg inhalation powder via DPI, once daily in the morning. Subjects may receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/VI (100/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)
- FF/VI (200/25) mcg dual combination therapy (Active Comparator): Subjects will receive FF/VI (200/25) mcg inhalation powder via DPI, once daily in the morning. Subjects may receive albuterol/salbutamol as a rescue medication when needed during the treatment period.
  Interventions: Drug: FF/VI (100/25) mcg; Drug: FF/VI (200/25) mcg; Drug: Fluticasone/salmeterol (FSC); Drug: Albuterol/salbutamol; Device: ELLIPTA DPI; Device: DISKUS DPI; Device: METERED-DOSE INHALER (MDI)

INTERVENTIONS:
Drug: FF/UMEC/VI (100/31.25/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation once-daily [QD] in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 100 mcg in each blister and the second strip contains UMEC 31.25 mcg and VI 25 mcg in each blister.
  Arms: FF/UMEC/VI (100/31.25/25) mcg closed triple therapy
Drug: FF/UMEC/VI (100/62.5/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation, QD in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 100 mcg in each blister and the second strip contains UMEC 62.5 mcg and VI 25 mcg in each blister.
  Arms: FF/UMEC/VI (100/62.5/25) mcg closed triple therapy
Drug: FF/UMEC/VI (200/31.25/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation, QD in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 200 mcg in each blister and the second strip contains UMEC 31.25 mcg and VI 25 mcg in each blister.
  Arms: FF/UMEC/VI (200/31.25/25) mcg closed triple therapy
Drug: FF/UMEC/VI (200/62.5/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation, QD in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 200 mcg in each blister and the second strip contains UMEC 62.5 mcg and VI 25 mcg in each blister.
  Arms: FF/UMEC/VI (200/62.5/25) mcg closed triple therapy
Drug: FF/VI (100/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation, QD in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 100 mcg in each blister and the second strip contains VI 25 mcg in each blister.
Drug: FF/VI (200/25) mcg — Dry white powder delivered via the ELLIPTA DPI (one inhalation, QD in the morning). The ELLIPTA DPI holds 2 individual blister strips with 30 blisters on each strip: the first strip contains FF 200 mcg in each blister and the second strip contains VI 25 mcg in each blister.
  Arms: FF/VI (200/25) mcg dual combination therapy
Drug: Fluticasone/salmeterol (FSC) — Dry white powder delivered via the DISKUS DPI (one inhalation twice daily: one in the morning and one in the evening). The DISKUS DPI holds a strip of 60 blisters; each blister contains FP 250 mcg and 50 mcg of salmeterol.
Drug: Albuterol/salbutamol — This is a rescue medication administered via metered-dose inhaler (MDI) which will be used when needed during the study.
Device: ELLIPTA DPI — The ELLIPTA device will be used during the stabilization period and the treatment period. The ELLIPTA DPI is a moulded plastic two-sided device that can hold two individual blister strips which contain powder formulation for oral inhalation.
Device: DISKUS DPI — The DISKUS device will be used during the run-in period. The DISKUS DPI is a plastic inhalation delivery system containing a single-foil blister strip of a powder formulation of FSC for oral inhalation.
Device: METERED-DOSE INHALER (MDI) — Albuterol/salbutamol (rescue medication) will be delivered via metered-dose inhaler (MDI) will be used for reversibility testing.

SUMMARY:
A once-daily 'closed' triple FDC therapy of FF/UMEC/VI via a single ELLIPTA® dry powder inhaler (DPI) is being developed by GlaxoSmithKline (GSK) with the aim of providing a new treatment option for the management of asthma by improving lung function, health-related quality of life (HRQoL) and symptom control over established combination therapies. This is a phase III, multi-center, active-controlled, double-blind, parallel-group study to compare the efficacy, safety and tolerability of the FDC of FF/UMEC/VI with the FDC of FF/VI. This study has 5 phases: Pre-Screening (Visit 0), Screening/Run-in, Enrolment/Stabilization, Randomization/Treatment, and Follow up. At Visit 1 (Screening), subjects meeting all protocol defined inclusion/exclusion criteria will enter a 3-week run-in period and will receive fixed dose inhaled corticosteroid/long-acting beta agonist (ICS/LABA) (fluticasone/salmeterol, 250/50 micrograms (mcg), via the DISKUS® DPI) one inhalation twice a day. At Visit 2 (Enrolment), eligible subjects will be enrolled into the 2-week stabilization period to receive FF/VI (100/25 mcg via the ELLIPTA DPI once a day, in the morning). At the conclusion of the stabilization period (Visit 3), all subjects who meet the pre-defined randomization criteria will be randomized 1:1:1:1:1:1 during the treatment period to receive either FF/UMEC/VI (100/62.5/25 mcg; 200/62.5/25 mcg; 100/31.25/25 mcg; 200/31.25/25 mcg) or FF/VI (100/25 mcg; 200/25 mcg) via the ELLIPTA DPI once daily in the morning. The duration of the treatment period is variable but will be a minimum of 24 weeks and a maximum of 52 weeks. Subjects will have up to 6 on-treatment clinic visits scheduled at Visits 3, 4, 5, 6, 7 and 8/End of Study (EOS) (Weeks 0, 4, 12, 24, 36 and 52, respectively). A follow-up visit will be conducted approximately 7 days after the end of treatment period or, if applicable, after the early withdrawal visit. Subjects will be provided with short acting albuterol/salbutamol to be used on an as-needed basis (rescue medication) throughout the study. Approximately 2250 subjects will be randomized, with approximately 375 subjects randomized to each of the 6 double-blind treatment arms to ensure approximately 337 evaluable subjects per treatment arm. DISKUS and ELLIPTA are registered trademarks of GSK groups of companies.

ELIGIBILITY:
Inclusion Criteria for Screening

* Age: 18 years of age or older at the time of signing the informed consent.
* Diagnosis: Subjects with a diagnosis of asthma as defined by the National Institutes of Health at least one year prior to Visit 0.
* Symptomatic: Subjects with inadequately controlled asthma (ACQ-6 score >=1.5) despite ICS/LABA maintenance therapy at Visit 1.
* Asthma Control: In the 1 year prior to Visit 1

  * A documented healthcare contact for acute asthma symptoms or
  * A documented temporary change in asthma therapy for acute asthma symptoms, according to a pre-specified asthma action plan (or equivalent)
* Current Asthma Maintenance Therapy: Subjects are eligible if they have required daily ICS/LABA for at least 12 weeks prior to Visit 0 with no changes to maintenance asthma medications during the 6 weeks immediately prior to Visit 0 (including no changes to a stable total dose of ICS of >250 mcg/day fluticasone proprionate [FP, or equivalent]).
* Spirometry: A best pre-bronchodilator morning (ante meridian [AM]) FEV1 >=30% and <85% of the predicted normal value at Visit 1. Predicted values will be based upon the European Respiratory Society (ERS) Global Lung Function Initiative.
* Reversibility of Disease: airway reversibility defined as >=12% and >=200 milliliter (mL) increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol at Visit 1.
* If the subject does not meet the above reversibility criteria at Visit 1 then the reversibility assessment may be repeated once within 7 days of Visit 1 if either criteria a) or b) are met: a) >=9% increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol at Visit 1. b) Documented evidence of a reversibility assessment within 1 year prior to Visit 1 which demonstrated a post-bronchodilator increase in FEV1 of >=12% and >=200 mL.

Should the subject successfully demonstrate airway reversibility (defined as >=12% and >=200 mL increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol) at the second attempt then, provided that all other eligibility criteria assessed at Visit 1 are met, the subject may enter the 3-week run-in period.

* Short-Acting beta2 Agonists (SABAs): All subjects must be able to replace their current SABA inhaler with albuterol/salbutamol aerosol inhaler at Visit 1 as needed for the duration of the study. Subjects must be judged capable of withholding albuterol/salbutamol for at least 6 hours prior to study visits.
* Male or eligible Female, defined as having documentation of non-reproductive potential or reproductive potential as follows:

A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test), not lactating, is not planning on becoming pregnant during the study and at least one of the following conditions applies: Non-reproductive potential defined as pre-menopausal females with documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or hysterectomy or documented bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea with an appropriate clinical profile (e.g., age appropriate, >45 years, in the absence of hormone replacement therapy). In questionable cases for women <60 years of age, a blood sample with simultaneous follicle stimulating hormone and estradiol falling into the central laboratory's postmenopausal reference range is confirmatory. Females under 60 years of age, who are on hormone replacement therapy (HRT) and whose menopausal status is in doubt, are required to use a highly effective method to avoid pregnancy if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, subjects can resume use of HRT during the study without use of a highly effective method to avoid pregnancy; Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from the screening visit until after the last dose of study medication and completion of the follow-up visit. The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form and in this protocol. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.

Exclusion Criteria for Screening

* Pneumonia: Chest X-ray documented pneumonia in the 6 weeks prior to Visit 1.
* Asthma Exacerbation: Any asthma exacerbation requiring a change in maintenance asthma therapy in the 6 weeks prior to Visit 1. Note: Subjects requiring a temporary change in asthma therapy (e.g., oral corticosteroids or increased dose of ICS) to treat an exacerbation in the 6 weeks prior to Visit 1 are not explicitly excluded at Visit 1 provided that, at the Investigator's discretion, the subject's condition is stable after they have resumed their pre-exacerbation maintenance asthma therapy (without modification) and they are considered appropriate for enrolment into this study of up to 12 month's duration.
* Chronic Obstructive Pulmonary Disease: Subjects with the diagnosis of chronic obstructive pulmonary disease, as per Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, including history of exposure to risk factors (i.e., especially tobacco smoke, occupational dusts and chemicals, smoke from home cooking and heating fuels) and a post-albuterol/salbutamol FEV1/Forced Vital Capacity (FVC) ratio of <0.70 and a post-albuterol/salbutamol FEV1 of =<70% of predicted normal values and onset of disease >=40 years of age.
* Concurrent respiratory disorders: Subjects with current evidence of pneumonia, active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases or abnormalities other than asthma.
* Risk Factors for Pneumonia: Immune suppression (e.g., human immunodeficiency virus, Lupus) or other risk factors for pneumonia (e.g., neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis).
* Patients at potentially high risk (e.g., very low body mass index (BMI), severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator.
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria.
* Clinically significant Electrocardiogram abnormality: Evidence of a clinically significant abnormality in the 12-lead ECG performed during screening. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: Atrial fibrillation (AF) with rapid ventricular rate >120 Beats Per Minute (BPM); sustained or non-sustained ventricular tachycardia (VT); Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 milliseconds (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.
* Unstable or life threatening cardiac disease: Subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure.
* Antimuscarinic effects: Subjects with a medical condition such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction should only be included if in the opinion of the Investigator the benefit outweighs the risk and that the condition would not contraindicate study participation.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol for the 6-hour period required prior to spirometry testing at each study visit.
* Tobacco Use: Subjects who are: Current smokers (defined as subjects who have used inhaled tobacco products within the 12 months prior to Visit 1 [i.e., cigarettes, e-cigarettes/vaping, cigars or pipe tobacco]) or former smokers with a smoking history of >=10 pack years (e.g., >=20 cigarettes/day for 10 years).
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Allergy or Hypersensitivity: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Affiliation with Investigator site: Study Investigators, sub-Investigators, study coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.

Inclusion Criteria for Enrolment

* Inadequately controlled asthma: Subjects with inadequately controlled asthma (ACQ-6 score >=1.5) at Visit 2.
* Percent-predicted FEV1: A best pre-bronchodilator morning (AM) FEV1 >=30% and <90% of the predicted normal value at Visit 2. Predicted values will be based upon the ERS Global Lung Function Initiative
* Liver function tests at Visit 1: alanine aminotransferase (ALT) <2 x upper limit of normal (ULN); alkaline phosphatase <=1.5xULN; bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Compliance with completion of the Daily eDiary reporting defined as completion of all questions/assessments on >=4 of the last 7 days during the run-in period.

Exclusion Criteria for Enrolment

* Respiratory Infection: Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Severe asthma exacerbation: Evidence of a severe exacerbation during screening or the run-in period, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Asthma medication: Changes in asthma medication (excluding run-in medication and albuterol/salbutamol inhalation aerosol provided at Visit 1).
* Laboratory test abnormalities: Evidence of clinically significant abnormal laboratory tests during screening or run-in which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality.

Inclusion Criteria for Randomization

* Compliance with completion of the Daily eDiary reporting defined as completion of all questions/assessments on >=4 of the last 7 days during the stabilization period.

Exclusion Criteria for Randomization

* Respiratory Infection: Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the stabilization period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Severe asthma exacerbation: Evidence of a severe exacerbation during enrolment or the stabilization period, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an inpatient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Asthma medication: Changes in asthma medication (excluding stabilization period medication provided at Visit 2 and albuterol/salbutamol inhalation aerosol provided at Visit 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2436 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (295):
- United States (92):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Canton, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Escondico, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Lafayette, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocoee, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Michigan City, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Rochester, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Hendersonville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Lampasas, Texas
  - GSK Investigational Site, Live Oak, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, Missouri City, Texas
  - GSK Investigational Site, Pharr, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Seattle, Washington
- Argentina (13):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Paraná, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Australia (9):
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Golden Beach
- Canada (16):
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Victoriaville, Quebec
  - GSK Investigational Site, Québec
- Germany (13):
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (11):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Civitanova Marche (MC), The Marches
  - GSK Investigational Site, Pisa, Tuscany
- Japan (30):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shimane
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamaguchi
  - GSK Investigational Site, Yamanashi
- Netherlands (9):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Poland (15):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Kościan
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Zgierz
- Romania (14):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Slobozia
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Târgu Mureş
  - GSK Investigational Site, Timișoara
- Russia (27):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Khantymansiysk
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Ulan-Ude
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (11):
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Pretoria West
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Tygerberg
- South Korea (8):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Cheongju-si, Chungcheongbuk-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
  - GSK Investigational Site, Wonju-si, Kanwon-do
- Spain (15):
  - GSK Investigational Site, Alcobendas, Madrid
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, Girona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Las Palmas
  - GSK Investigational Site, Loja/ Granada
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Zaragoza
- United Kingdom (12):
  - GSK Investigational Site, Aberdeen, Aberdeenshire
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Wishaw, Lanarkshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Corby, Northamptonshire
  - GSK Investigational Site, Bexhill-on-Sea, Sussex East
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Edgbaston
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Sidcup, Kent
  - GSK Investigational Site, Trowbridge

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20767

REFERENCES:
- [Derived] Oppenheimer J, Pavord ID, Corbridge T, Crawford J, Gould S, Hamouda M, Howarth P, Burrows E, Moore A, Noorduyn SG, Slade D, Weng S, Lugogo N. Evaluating Asthma Clinical Remission with Inhaled Therapy: Post Hoc Analyses of CAPTAIN. Adv Ther. 2025 Dec 24. doi: 10.1007/s12325-025-03442-x. Online ahead of print. PMID 41442024
- [Derived] Oppenheimer J, Hanania NA, Chaudhuri R, Sagara H, Bailes Z, Fowler A, Peachey G, Pizzichini E, Slade D. Clinic vs Home Spirometry for Monitoring Lung Function in Patients With Asthma. Chest. 2023 Nov;164(5):1087-1096. doi: 10.1016/j.chest.2023.06.029. Epub 2023 Jun 27. PMID 37385337
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Nakamura Y, Hozawa S, Sagara H, Ohbayashi H, Lee LA, Crawford J, Tamaoki J, Nishi T, Fowler A. Efficacy and safety of once-daily, single-inhaler fluticasone furoate/umeclidinium/vilanterol versus fluticasone furoate/vilanterol in Japanese patients with inadequately controlled asthma: the CAPTAIN study. Curr Med Res Opin. 2021 Sep;37(9):1657-1665. doi: 10.1080/03007995.2021.1944849. Epub 2021 Jul 14. PMID 34162298
- [Derived] Yang S, Lee LA, Sule N, Fowler A, Peachey G. Population Pharmacokinetic Modeling of Fluticasone Furoate, Umeclidinium Bromide, and Vilanterol in Patients with Asthma, Using Data from a Phase IIIA Study (CAPTAIN). Clin Pharmacokinet. 2021 Jul;60(7):887-896. doi: 10.1007/s40262-021-00988-1. Epub 2021 Feb 18. PMID 33598874
- [Derived] Lee LA, Bailes Z, Barnes N, Boulet LP, Edwards D, Fowler A, Hanania NA, Kerstjens HAM, Kerwin E, Nathan R, Oppenheimer J, Papi A, Pascoe S, Brusselle G, Peachey G, Sule N, Tabberer M, Pavord ID. Efficacy and safety of once-daily single-inhaler triple therapy (FF/UMEC/VI) versus FF/VI in patients with inadequately controlled asthma (CAPTAIN): a double-blind, randomised, phase 3A trial. Lancet Respir Med. 2021 Jan;9(1):69-84. doi: 10.1016/S2213-2600(20)30389-1. Epub 2020 Sep 9. PMID 32918892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 322 centers across 15 countries.
Pre-assignment Details: Total 5185 participants were screened and 2436 participants were enrolled into the study and received the study treatment.
Groups:
- FF/VI 100/25 mcg: Participants received Fluticasone Furoate/ Vilanterol (FF/VI) 100/25 micrograms (mcg) inhalation powder via dry powder inhaler (DPI), once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI 100/ 31.25/25 mcg: Participants received Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) 100/31.25/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI 100/62.5/25 mcg: Participants received FF/UMEC/VI 100/62.5/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/VI 200/25 mcg: Participants received FF/VI 200/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI 200/ 31.25/25 mcg: Participants received FF/UMEC/VI 200/31.25/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI 200/62.5/25 mcg: Participants received FF/UMEC/VI 200/62.5/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
Period: Overall Study
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Started | 407 | 405 | 406 | 406 | 404 | 408
Completed | 374 | 374 | 383 | 378 | 381 | 384
Not Completed | 33 | 31 | 23 | 28 | 23 | 24
Not completed — Adverse Event | 9 | 3 | 2 | 2 | 3 | 2
Not completed — Lack of Efficacy | 2 | 3 | 4 | 2 | 1 | 1
Not completed — Protocol Violation | 3 | 7 | 5 | 6 | 2 | 2
Not completed — Protocol defined withdrawal criteria met | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 4 | 2 | 4 | 2 | 4
Not completed — Physician Decision | 2 | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 14 | 13 | 9 | 12 | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg | Total
Number analyzed (Participants) | 407 | 405 | 406 | 406 | 404 | 408 | 2436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (13.03) | 51.7 (13.27) | 52.9 (13.39) | 53.9 (13.30) | 53.5 (13.12) | 53.7 (12.50) | 53.2 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 262 | 248 | 252 | 240 | 258 | 1514
  Male | 153 | 143 | 158 | 154 | 164 | 150 | 922
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American (AA) | 20 | 21 | 17 | 26 | 11 | 24 | 119
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Race: Asian-Central/South Asian Heritage (H.) | 5 | 4 | 1 | 5 | 9 | 0 | 24
  Race: Asian-Japanese H./East Asian H./SouthEast Asian H. | 54 | 55 | 50 | 53 | 55 | 52 | 319
  Race: Mixed Asian Race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Race: White | 326 | 319 | 338 | 316 | 325 | 326 | 1950
  Race: American Indian or Alaska Native and Black or AA | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: American Indian or Alaska Native and White | 1 | 0 | 0 | 0 | 0 | 2 | 3
  Race: Asian and Black or African American and White | 0 | 1 | 0 | 2 | 0 | 0 | 3
  Race: Asian and White | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: Black or African American and White | 1 | 2 | 0 | 3 | 0 | 1 | 7
  Race: Missing | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal volume of air that can be forcefully exhaled in one second. Trough FEV1 on treatment is defined as the highest FEV1 value obtained prior to the morning dose of investigational product. Baseline value is the last acceptable/borderline acceptable pre-dose FEV1 prior to randomized treatment start date (pre-dose at Day 1). Change from Baseline value is the value at Week 24 minus the Baseline value. Intent-to-Treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error, who did not receive the study drug. Treatment policy estimand was assessed, including all on- and post-treatment data. Different participants may have been analyzed at different time points; thus, overall number of participants analyzed reflects everyone in ITT Population without missing covariate information, with Baseline and at least one post-baseline measurement. Mixed Model Repeated Measures(MMRM) was used.
Time Frame: Baseline (pre-dose at Day 1) and Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed. Participants with Baseline value and at least one post-baseline measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 400 | 399 | 404 | 403 | 399 | 405
Liters | 0.024 (0.0157) | 0.120 (0.0157) | 0.134 (0.0155) | 0.076 (0.0156) | 0.157 (0.0156) | 0.168 (0.0155)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/ 31.25/25 mcg; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — p-value was calculated using MMRM with covariates of treatment, age, sex, region, Baseline value, pre-study inhaled corticosteroids (ICS) dosage at screening, and visit, interaction terms for Baseline value by visit and treatment by visit; Least Squares Mean Difference = 0.096, 95% CI 2-sided [0.052 to 0.139], Standard Error of Mean 0.0222
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/62.5/25 mcg; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — p-value was calculated using MMRM with covariates of treatment, age, sex, region, Baseline value, pre-study ICS dosage at screening, and visit, interaction terms for Baseline value by visit and treatment by visit; Least Squares Mean Difference = 0.110, 95% CI 2-sided [0.066 to 0.153], Standard Error of Mean 0.0221
Statistical Analysis 3: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/ 31.25/25 mcg; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.082, 95% CI 2-sided [0.039 to 0.125], Standard Error of Mean 0.0221
Statistical Analysis 4: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/62.5/25 mcg; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.092, 95% CI 2-sided [0.049 to 0.135], Standard Error of Mean 0.0220

2. Secondary Outcome: Annualized Rate of Moderate and Severe Asthma Exacerbations
Description: A moderate asthma exacerbation is considered to be a deterioration in asthma symptoms or in lung function, or increased rescue bronchodilator use lasting for at least 2 days or more, but not be severe enough to warrant systemic corticosteroid use (or a doubling or more of the maintenance systemic corticosteroid dose, if applicable) for 3 days or more and/or hospitalization. It is an event that, when recognized, should result in a temporary change in treatment, to prevent it from becoming severe. A severe asthma exacerbation is defined as the deterioration of asthma requiring the use of systemic corticosteroids (tablets,suspension or injection), or an increase from a stable maintenance dose (For participants receiving maintenance systemic corticosteroids, at least double the maintenance systemic corticosteroid dose for at least 3 days is required), for at least 3 days or an inpatient hospitalization or emergency department visit because of asthma, requiring systemic corticosteroids.
Time Frame: Up to Week 52
Population: ITT Population. Only participants with at least one day on study post-randomization were analyzed. Analysis used pooled data from two FF/UMEC/VI arms for each fixed UMEC dose compared to pooled data from two FF/VI arms to provide a more precise estimate for the treatment effect of the addition of UMEC to FF/VI.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Groups:
- FF/VI: Participants received FF/VI 100/25 mcg or 200/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI (UMEC 31.25 mcg): Participants received FF/UMEC/VI 100/31.25/25 mcg or 200/31.25/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
- FF/UMEC/VI (UMEC 62.5 mcg): Participants received FF/UMEC/VI 100/62.5/25 mcg or 200/62.5/25 mcg inhalation powder via DPI, once daily in the morning up to 52 weeks. Participants were allowed to take albuterol/salbutamol as a rescue medication when needed during the treatment period.
Arm/Group | FF/VI | FF/UMEC/VI (UMEC 31.25 mcg) | FF/UMEC/VI (UMEC 62.5 mcg)
Number analyzed (Participants) | 813 | 809 | 814
Exacerbations per year | 0.70 [0.61 to 0.80] | 0.68 [0.60 to 0.78] | 0.61 [0.53 to 0.70]
Statistical Analysis 1: Comparison: FF/VI vs FF/UMEC/VI (UMEC 31.25 mcg); Test type: Superiority; p = 0.778, Negative Binomial Model — p-value was calculated using Generalized linear model with covariates for age, sex, region, treatment group, stratification by pre-study ICS dosage at screening, and severe asthma exacerbations in the previous year (0, 1, >=2); Rate Ratio = 0.97, 95% CI 2-sided [0.81 to 1.17] — Treatment policy estimand was assessed, including all on- and post-treatment data
Statistical Analysis 2: Comparison: FF/VI vs FF/UMEC/VI (UMEC 62.5 mcg); Test type: Superiority; p = 0.151, Negative Binomial Model — [p-value comment as in outcome 2, analysis 1]; Rate Ratio = 0.87, 95% CI 2-sided [0.72 to 1.05] — Treatment policy estimand was assessed, including all on- and post-treatment data

3. Secondary Outcome: Mean Change From Baseline in Clinic FEV1 at 3 Hours Post Study Treatment at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal volume of air that can be forcefully exhaled in one second. Baseline value is the last acceptable/borderline acceptable pre-dose FEV1 prior to randomized treatment start date (pre-dose at Day 1). Change from Baseline value is the value at Week 24 (recorded at 3 hours post dose) minus the Baseline value.
Time Frame: Baseline (pre-dose at Day 1) and 3 hours post dose at Week 24
Population: ITT Population. Only those participants with available Baseline and on-treatment data at Week 24 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 369 | 375 | 379 | 377 | 371 | 378
Liters | 0.132 (0.0160) | 0.220 (0.0159) | 0.243 (0.0158) | 0.168 (0.0159) | 0.256 (0.0160) | 0.286 (0.0158)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/ 31.25/25 mcg; Test type: Superiority; p < 0.001, ANCOVA — p-value was calculated using Analysis of Covariance (ANCOVA) with covariates of treatment, age, sex, region, Baseline value, and pre-study ICS dosage at screening; Least Squares Mean Difference = 0.088, 95% CI 2-sided [0.044 to 0.132], Standard Error of Mean 0.0226
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/62.5/25 mcg; Test type: Superiority; p < 0.001, ANCOVA — p-value was calculated using ANCOVA with covariates of treatment, age, sex, region, Baseline value, and pre-study ICS dosage at screening; Least Squares Mean Difference = 0.111, 95% CI 2-sided [0.067 to 0.155], Standard Error of Mean 0.0225
Statistical Analysis 3: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/ 31.25/25 mcg; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Least Squares Mean Difference = 0.088, 95% CI 2-sided [0.044 to 0.132], Standard Error of Mean 0.0225
Statistical Analysis 4: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/62.5/25 mcg; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 2]; Least Squares Mean Difference = 0.118, 95% CI 2-sided [0.074 to 0.162], Standard Error of Mean 0.0224

4. Secondary Outcome: Mean Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) Total Score at Week 24
Description: The ACQ-7 consists of 7 attributes of asthma control, of which 6 to be self-completed by participant in a 6-item questionnaire, enquire about frequency and/or severity of symptoms over the previous week on: nocturnal awakening, symptoms on waking in the morning, activity limitation, shortness of breath, wheeze, and rescue medication use. The seventh attribute measures the lung function, which was included via pre-bronchodilator FEV1 % predicted value. All 7 items of ACQ have response on 0-6 ordinal scale (0=no impairment/limitation, 6=total impairment/limitation). The total score is calculated as the average of all non-missing item responses, ranges from 0 to 6. Higher score indicates worst symptoms. Treatment policy estimand was assessed, including all on- and post-treatment data. Baseline value was at randomization visit (pre-dose,Day 1). Change from Baseline was defined as value at Week 24 minus Baseline value.
Time Frame: Baseline (pre-dose at Day 1) and Week 24
Population: ITT Population. Participants with available data at Baseline and at least one time point post-baseline were analyzed. Analysis used pooled data from two FF/UMEC/VI arms for each fixed UMEC dose compared to pooled data from two FF/VI arms to provide a more precise estimate for the treatment effect of the addition of UMEC to FF/VI.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/VI | FF/UMEC/VI (UMEC 31.25 mcg) | FF/UMEC/VI (UMEC 62.5 mcg)
Number analyzed (Participants) | 784 | 784 | 790
Scores on a scale | -0.678 (0.0240) | -0.734 (0.0240) | -0.767 (0.0238)
Statistical Analysis 1: Comparison: FF/VI vs FF/UMEC/VI (UMEC 31.25 mcg); Test type: Superiority; p = 0.094, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.057, 95% CI 2-sided [-0.124 to 0.010], Standard Error of Mean 0.0340
Statistical Analysis 2: Comparison: FF/VI vs FF/UMEC/VI (UMEC 62.5 mcg); Test type: Superiority; p = 0.008, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.089, 95% CI 2-sided [-0.156 to -0.023], Standard Error of Mean 0.0338

5. Secondary Outcome: Mean Change From Baseline in Saint George's Respiratory Questionnaire (SGRQ) Total Score at Week 24
Description: The SGRQ had 50 questions (scored from 0 to 100 where 0 indicates best and 100 indicates worst health) designed to measure quality of life (QoL) of participants with airway obstruction, measuring symptoms, impact, and activity. The questions are designed to be self-completed by the participant with a recall over the past 3 months. SGRQ total score was calculated by summing the pre-assigned weights of answers, dividing by the sum of the maximum weights for items in SGRQ and multiplying by 100. SGRQ total score ranges from 0 to 100 where 0 indicates best and 100 indicates worst health. A change of 4 points is considered a clinically relevant change. Treatment policy estimand was assessed, including all on- and post-treatment data. Baseline value was at randomization visit (pre-dose at Day 1). Change from Baseline value is the value at Week 24 minus the Baseline value.
Time Frame: Baseline (pre-dose at Day 1) and Week 24
Population: ITT Population. Participants with a Baseline value and at least one post-baseline measurement were analyzed. Analysis used pooled data from two FF/UMEC/VI arms for each fixed UMEC dose compared to pooled data from two FF/VI arms to provide a more precise estimate for the treatment effect of the addition of UMEC to FF/VI.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/VI | FF/UMEC/VI (UMEC 31.25 mcg) | FF/UMEC/VI (UMEC 62.5 mcg)
Number analyzed (Participants) | 784 | 782 | 795
Scores on a scale | -11.39 (0.491) | -10.29 (0.494) | -11.69 (0.487)
Statistical Analysis 1: Comparison: FF/VI vs FF/UMEC/VI (UMEC 31.25 mcg); Test type: Other; p = 0.115, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 1.10, 95% CI 2-sided [-0.27 to 2.47], Standard Error of Mean 0.697
Statistical Analysis 2: Comparison: FF/VI vs FF/UMEC/VI (UMEC 62.5 mcg); Test type: Other; p = 0.662, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-1.66 to 1.05], Standard Error of Mean 0.692

6. Secondary Outcome: Mean Change From Baseline in Evaluating Respiratory Symptoms (E-RS) Total Score Over Weeks 21 to 24 (Inclusive) of the Treatment Period
Description: The E-RS in Chronic Obstructive Pulmonary Disease (COPD) consists of 11 items. E-RS captures information related to respiratory symptoms, i.e. breathlessness, cough, sputum production, chest congestion and chest tightness. The E-RS was completed daily and data was derived by 4-weekly intervals, requiring at least 50% of data to be present during a period. 7 items are scored from 0 (not at all) to 4 (extreme) and 4 items are scored from 0 (not at all) to 3 (extreme). The E-RS total score was calculated by taking sum of all the items. The E-RS total score has a scoring range of 0 to 40, with higher scores indicating more severe respiratory symptoms. Treatment policy estimand was assessed, including all on- and post-treatment data. Baseline value was the mean value of 14 days prior to randomization. Change from Baseline was calculated as post-baseline value (mean of daily E-RS total scores during Week 21 to 24 ) minus Baseline value.
Time Frame: Baseline (14 days prior to randomization) and Weeks 21 to 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/VI | FF/UMEC/VI (UMEC 31.25 mcg) | FF/UMEC/VI (UMEC 62.5 mcg)
Number analyzed (Participants) | 787 | 796 | 802
Scores on a scale | -2.47 (0.131) | -2.60 (0.130) | -2.89 (0.130)
Statistical Analysis 1: Comparison: FF/VI vs FF/UMEC/VI (UMEC 31.25 mcg); Test type: Other; p = 0.479, Mixed Model Repeated Measures — p-value was calculated using MMRM with covariates of treatment, age, sex, region, Baseline value, pre-study ICS dosage at screening, and 4-weekly period, interaction terms for Baseline value by 4-weekly period and treatment by 4-weekly period; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.49 to 0.23], Standard Error of Mean 0.185
Statistical Analysis 2: Comparison: FF/VI vs FF/UMEC/VI (UMEC 62.5 mcg); Test type: Other; p = 0.023, Mixed Model Repeated Measures — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.42, 95% CI 2-sided [-0.78 to -0.06], Standard Error of Mean 0.184

7. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Common (>=3%) Non-SAE
Description: Adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, events associated with liver injury and impaired liver function, or any other situation according to medical or scientific judgment were categorized as SAE. Number of participants with any SAE and common (>=3%) non-SAEs are presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 407 | 405 | 406 | 406 | 404 | 408
Participants
  Common non-SAE | 136 | 150 | 135 | 122 | 127 | 122
  SAE | 25 | 18 | 23 | 21 | 23 | 21

8. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were performed during the study using an automated ECG machine. All ECG measurements were made with the participant in a supine position having rested in this position for approximately 5 minutes before each reading. The number of participants with worst case post-Baseline abnormal ECG findings were reported.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 401 | 398 | 398 | 397 | 399 | 404
Participants | 115 | 118 | 109 | 109 | 106 | 108

9. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 24
Description: Blood pressure (systolic and diastolic) was measured in the sitting position after approximately 5 minutes rest. Baseline value is the last acceptable/borderline acceptable value prior to randomized treatment start date (pre-dose at Day 1). Change from Baseline value is the value at the clinic visit minus the Baseline value. Different participants may have been analyzed at different time points; thus, overall number of participants analyzed reflects everyone in ITT Population without missing covariate information, with Baseline and at least one post-baseline measurement.
Time Frame: Baseline (pre-dose at Day 1) and Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed. Participants with a Baseline value and at least one post-baseline measurement were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 401 | 398 | 399 | 397 | 399 | 402
Millimeter of mercury
  SBP | 1.6 (0.53) | 0.6 (0.53) | 1.1 (0.52) | 0.2 (0.53) | 0.8 (0.53) | 0.9 (0.52)
  DBP | 0.4 (0.39) | 0.1 (0.39) | 1.3 (0.39) | 0.4 (0.39) | 0.2 (0.40) | 0.8 (0.39)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/ 31.25/25 mcg; Test type: Other; p = 0.172, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.5 to 0.4], Standard Error of Mean 0.75 — Comparison for SBP
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/62.5/25 mcg; Test type: Other; p = 0.436, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-2.0 to 0.9], Standard Error of Mean 0.74 — Comparison for SBP
Statistical Analysis 3: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/ 31.25/25 mcg; Test type: Other; p = 0.426, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.6, 95% CI 2-sided [-0.9 to 2.1], Standard Error of Mean 0.75 — Comparison for SBP
Statistical Analysis 4: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/62.5/25 mcg; Test type: Other; p = 0.349, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.7, 95% CI 2-sided [-0.8 to 2.2], Standard Error of Mean 0.74 — Comparison for SBP
Statistical Analysis 5: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/ 31.25/25 mcg; Test type: Other; p = 0.482, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-1.5 to 0.7], Standard Error of Mean 0.56 — Comparison for DBP
Statistical Analysis 6: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/62.5/25 mcg; Test type: Other; p = 0.142, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.8, 95% CI 2-sided [-0.3 to 1.9], Standard Error of Mean 0.56 — Comparison for DBP
Statistical Analysis 7: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/ 31.25/25 mcg; Test type: Other; p = 0.806, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-1.2 to 1.0], Standard Error of Mean 0.56 — Comparison for DBP
Statistical Analysis 8: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/62.5/25 mcg; Test type: Other; p = 0.447, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-0.7 to 1.5], Standard Error of Mean 0.55 — Comparison for DBP

10. Secondary Outcome: Mean Change From Baseline in Pulse Rate at Week 24
Description: Pulse Rate was measured in the sitting position after approximately 5 minutes rest. Baseline value is the last acceptable/borderline acceptable value prior to randomized treatment start date (pre-dose at Day 1). Change from Baseline value is the value at the clinic visit minus the Baseline value. Different participants may have been analyzed at different time points; thus, overall number of participants analyzed reflects everyone in ITT Population without missing covariate information, with Baseline and at least one post-baseline measurement.
Time Frame: Baseline (pre-dose at Day 1) and Week 24
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 401 | 398 | 399 | 397 | 399 | 402
Beats per minute | -1.1 (0.43) | 0.2 (0.43) | -1.0 (0.43) | -0.7 (0.43) | -1.3 (0.44) | -0.5 (0.43)
Statistical Analysis 1: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/ 31.25/25 mcg; Test type: Other; p = 0.034, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 1.3, 95% CI 2-sided [0.1 to 2.5], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: FF/VI 100/25 mcg vs FF/UMEC/VI 100/62.5/25 mcg; Test type: Other; p = 0.839, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-1.1 to 1.3], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/ 31.25/25 mcg; Test type: Other; p = 0.349, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-1.8 to 0.6], Standard Error of Mean 0.61
Statistical Analysis 4: Comparison: FF/VI 200/25 mcg vs FF/UMEC/VI 200/62.5/25 mcg; Test type: Other; p = 0.768, Mixed Model Repeated Measures — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Difference = 0.2, 95% CI 2-sided [-1.0 to 1.4], Standard Error of Mean 0.61

11. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Values
Description: Blood samples were collected for assessment of clinical chemistry parameters, which included albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), direct bilirubin, total bilirubin, calcium, creatinine, glucose, potassium, protein, sodium and urea. Abnormal laboratory results are categorized as high or low with respect to their normal ranges. Participants having High and Low values from normal ranges for any parameter at any time post-baseline visits are presented.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 391 | 392 | 394 | 390 | 391 | 397
Participants
  Albumin, low | 2 | 0 | 0 | 1 | 0 | 0
  Albumin, high | 1 | 6 | 5 | 2 | 3 | 1
  ALT, low | 0 | 0 | 0 | 0 | 0 | 0
  ALT, high | 41 | 29 | 24 | 28 | 27 | 30
  AST, low | 0 | 0 | 0 | 0 | 0 | 0
  AST, high | 29 | 27 | 14 | 21 | 23 | 16
  ALP, low | 1 | 0 | 0 | 0 | 1 | 0
  ALP, high | 21 | 15 | 10 | 12 | 16 | 12
  Direct bilirubin, low | 0 | 0 | 0 | 0 | 0 | 0
  Direct bilirubin, high | 1 | 1 | 0 | 2 | 2 | 1
  Bilirubin, low | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, high | 9 | 12 | 5 | 15 | 17 | 13
  Calcium, low | 4 | 9 | 7 | 7 | 4 | 3
  Calcium, high | 4 | 12 | 10 | 11 | 8 | 7
  Creatinine, low | 54 | 62 | 49 | 63 | 60 | 64
  Creatinine, high | 7 | 7 | 8 | 6 | 9 | 8
  Glucose, low | 15 | 11 | 11 | 7 | 12 | 7
  Glucose, high | 74 | 71 | 70 | 76 | 66 | 73
  Potassium, low | 2 | 3 | 1 | 7 | 7 | 6
  Potassium, high | 15 | 13 | 11 | 9 | 12 | 19
  Protein, low | 3 | 0 | 5 | 3 | 1 | 2
  Protein, high | 0 | 1 | 3 | 2 | 3 | 1
  Sodium, low | 5 | 7 | 3 | 5 | 7 | 3
  Sodium, high | 6 | 7 | 7 | 4 | 5 | 7
  Urea, low | 3 | 4 | 5 | 3 | 3 | 1
  Urea, high | 13 | 17 | 3 | 11 | 11 | 13

12. Secondary Outcome: Number of Participants With Abnormal Hematology Values
Description: Blood samples were collected for assessment of hematology parameters, which included Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Platelets, Mean Corpuscular Hemoglobin (MCH) and Mean Corpuscular Volume (MCV). Abnormal laboratory results are categorized as high or low with respect to their normal ranges. Participants having High and Low values from normal ranges for any parameter at any time post-baseline visits are presented.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the specified time point were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
Number analyzed (Participants) | 391 | 390 | 392 | 391 | 391 | 397
Participants
  Basophils, low, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Basophils, low, n=390,390,391,389,389,396 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils, high, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Basophils, high, n=390,390,391,389,389,396 | 1 | 0 | 0 | 0 | 0 | 0
  Eosinophils, low, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Eosinophils, low, n=390,390,391,389,389,396 | 26 | 27 | 25 | 31 | 32 | 28
  Eosinophils, high, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Eosinophils, high, n=390,390,391,389,389,396 | 111 | 84 | 102 | 84 | 85 | 78
  Lymphocytes, low, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Lymphocytes, low, n=390,390,391,389,389,396 | 13 | 11 | 13 | 8 | 13 | 10
  Lymphocytes, high, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Lymphocytes, high, n=390,390,391,389,389,396 | 2 | 5 | 1 | 7 | 6 | 6
  Monocytes, low, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Monocytes, low, n=390,390,391,389,389,396 | 60 | 68 | 57 | 64 | 51 | 63
  Monocytes, high, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Monocytes, high, n=390,390,391,389,389,396 | 7 | 1 | 4 | 2 | 7 | 4
  Neutrophils, low, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Neutrophils, low, n=390,390,391,389,389,396 | 14 | 10 | 16 | 10 | 12 | 9
  Neutrophils, high, n=390,390,391,389,389,396: number analyzed (Participants) | 390 | 390 | 391 | 389 | 389 | 396
  Neutrophils, high, n=390,390,391,389,389,396 | 21 | 20 | 15 | 19 | 15 | 34
  Erythrocytes, low, n=391,390,392,391,391,397 | 14 | 16 | 11 | 15 | 21 | 22
  Erythrocytes, high, n=391,390,392,391,391,397 | 24 | 21 | 13 | 12 | 17 | 17
  Hematocrit, low, n=391,390,392,391,391,397 | 21 | 28 | 16 | 20 | 20 | 26
  Hematocrit, high, n=391,390,392,391,391,397 | 60 | 52 | 50 | 47 | 49 | 49
  Hemoglobin, low, n=391,390,392,391,391,397 | 32 | 47 | 40 | 40 | 37 | 34
  Hemoglobin, high, n=391,390,392,391,391,397 | 14 | 13 | 8 | 17 | 10 | 13
  Leukocytes, low, n=391,390,391,389,391,396: number analyzed (Participants) | 391 | 390 | 391 | 389 | 391 | 396
  Leukocytes, low, n=391,390,391,389,391,396 | 9 | 12 | 14 | 9 | 12 | 8
  Leukocytes, high, n=391,390,391,389,391,396: number analyzed (Participants) | 391 | 390 | 391 | 389 | 391 | 396
  Leukocytes, high, n=391,390,391,389,391,396 | 38 | 29 | 20 | 31 | 26 | 40
  Platelets, low, n=391,388,389,391,388,396: number analyzed (Participants) | 391 | 388 | 389 | 391 | 388 | 396
  Platelets, low, n=391,388,389,391,388,396 | 4 | 2 | 3 | 4 | 5 | 4
  Platelets, high, n=391,388,389,391,388,396: number analyzed (Participants) | 391 | 388 | 389 | 391 | 388 | 396
  Platelets, high, n=391,388,389,391,388,396 | 17 | 16 | 19 | 21 | 19 | 21
  MCH, low, n=391,390,392,391,391,397 | 40 | 47 | 24 | 34 | 41 | 25
  MCH, high, n=391,390,392,391,391,397 | 18 | 32 | 22 | 17 | 25 | 32
  MCV, low, n=391,390,392,391,391,397 | 20 | 22 | 10 | 15 | 19 | 14
  MCV, high, n=391,390,392,391,391,397 | 29 | 41 | 25 | 29 | 26 | 37

ADVERSE EVENTS:
Time Frame: Non-serious AEs and serious AEs were collected from start of study treatment (Week 0) up to Week 52
Description: Non-serious AEs and serious AEs were collected for ITT Population.
Arm/Group | FF/VI 100/25 mcg | FF/UMEC/VI 100/ 31.25/25 mcg | FF/UMEC/VI 100/62.5/25 mcg | FF/VI 200/25 mcg | FF/UMEC/VI 200/ 31.25/25 mcg | FF/UMEC/VI 200/62.5/25 mcg
All-Cause Mortality (participants affected / at risk) | 0/407 | 2/405 | 0/406 | 1/406 | 0/404 | 0/408
Serious Adverse Events (participants affected / at risk) | 25/407 | 18/405 | 23/406 | 21/406 | 23/404 | 21/408
Other Adverse Events (participants affected / at risk) | 136/407 | 150/405 | 135/406 | 122/406 | 127/404 | 122/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 mcg (N=407) | FF/UMEC/VI 100/ 31.25/25 mcg (N=405) | FF/UMEC/VI 100/62.5/25 mcg (N=406) | FF/VI 200/25 mcg (N=406) | FF/UMEC/VI 200/ 31.25/25 mcg (N=404) | FF/UMEC/VI 200/62.5/25 mcg (N=408)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 7 | 6 | 5 | 4
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 3 | 4 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 mcg (N=407) | FF/UMEC/VI 100/ 31.25/25 mcg (N=405) | FF/UMEC/VI 100/62.5/25 mcg (N=406) | FF/VI 200/25 mcg (N=406) | FF/UMEC/VI 200/ 31.25/25 mcg (N=404) | FF/UMEC/VI 200/62.5/25 mcg (N=408)
Nasopharyngitis (Infections and infestations) | 63 | 56 | 60 | 53 | 51 | 51
Upper respiratory tract infection (Infections and infestations) | 21 | 24 | 15 | 13 | 15 | 19
Bronchitis (Infections and infestations) | 14 | 18 | 15 | 19 | 16 | 22
Respiratory tract infection viral (Infections and infestations) | 11 | 17 | 10 | 7 | 12 | 9
Influenza (Infections and infestations) | 13 | 12 | 15 | 9 | 8 | 6
Pharyngitis (Infections and infestations) | 8 | 10 | 9 | 14 | 11 | 9
Headache (Nervous system disorders) | 30 | 31 | 36 | 23 | 27 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12 | 13 | 6 | 14 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02924688/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT02924688/SAP_001.pdf